CLINICAL TRIAL: NCT05361850
Title: Comparison of Deep Versus Awake Tracheal Extubation in Adults
Acronym: CDATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Navy (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Andrew Lee, Staff Anesthesiologist, United States Navy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMCP.2020.0097
Record Dates: First submitted 2022-04-23; First posted 2022-05-05 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Airway Complication of Anesthesia; Respiratory Complications of Care
Keywords: Awake Extubation; Deep Extubation
MeSH Terms: interventions — Airway Extubation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Awake Extubation (Active Comparator): Removal of the endotracheal tube while the patient is no longer under general anesthesia
  Interventions: Procedure: Extubation
- Deep Extubation (Active Comparator): Removal of the endotracheal tube while the patient is under general anesthesia
  Interventions: Procedure: Extubation

INTERVENTIONS:
Procedure: Extubation — Removal of the endotracheal tube

SUMMARY:
Prospective, randomized, single-blinded controlled study to compare the airway and respiratory complications of deep and awake tracheal extubations in adults.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status classification system for assessing the fitness of patients before surgery 1-3
* Meeting American Society of Anesthesiologists Practice Guidelines for Preoperative Fasting
* Adult patients age 18-64
* Favorable airway examinations (Mallampati 1 or 2, normal mouth opening, and intact neck extension)
* Scheduled cases in which tracheal intubation and general anesthesia are indicated

Exclusion Criteria:

* Patients with chronic obstructive pulmonary disease, pulmonary hypertension, interstitial lung disease, active respiratory infections, and/or uncontrolled asthma
* Unfavorable airway examinations (Mallampati 3 or 4, limited mouth opening, and/or inability to extend neck)
* Full stomach
* Known difficult intubation or mask ventilation
* Surgeries of the airway and intrathoracic surgeries
* Emergent surgeries
* Case duration >6 hours
* Pregnancy
* Patients scheduled to receive a protocolized anesthetic (Enhanced Recovery After Surgery aka ERAS)
* ASA Physical Status Classification 4 or 5
* Chronic diseases such as obstructive pulmonary disease, pulmonary hypertension, interstitial lung disease, active respiratory infections, and/or uncontrolled asthma
* Uncontrolled gastroesophageal reflux disease (heartburn) defined by presence of symptoms despite compliance with appropriate medication regimen
* Patient scheduled to receive a protocolized anesthetic ie Enhanced Recovery After Anesthesia (ERAS)
* Surgeries requiring prone positioning

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Aggregate Rate of Airway and Respiratory Complications | Peri-extubation period
  Coughing, obstruction, apnea, hypoxemia, bronchospasm, laryngospasm, aspiration

SECONDARY OUTCOMES:
Incidence and Severity of Postoperative Sore Throat | At time of transfer from PACU Phase 1 to PACU Phase 2 once PACU Phase 1 discharge criteria met, minimum of twenty minutes
  Sore Throat Rated on 0-10 Visual Analog Scale
Peri-extubation Heart Rate | Peri-extubation period
  Beats per minute, Incidence and Severity of Tachycardia (defined as 20% from Baseline Heart Rate)
Peri-extubation Blood Pressure | Peri-extubation period
  Systolic, Diastolic, and Mean Arterial Pressure in Millimeters of Mercury by Non-Invasive Blood Pressure, Incidence and Severity of Hypertension and Hypotension (defined as 20% from Baseline Blood Pressure)
End-of-Surgery to Out-Of-Room Time | From End-of-Surgery Time (defined by surgical dressing application) to Out-of-Room Time (defined by patient physically leaving operating room), up to two hours
  Duration in Minutes
Peri-extubation Agitation | From ten minutes prior to extubation to transfer time from PACU Phase 1 to PACU Phase 2 (minimum PACU Phase 1 stay 20 minutes)
  Incidence of Richmond Agitation-Sedation Scale score >=2

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center Portsmouth, Portsmouth, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee MA, Schenke PW, Faller MR, DeYoung HR, Adams AR. A comparison of deep versus awake tracheal extubation in adults: a randomized controlled trial. BMC Anesthesiol. 2025 Jul 31;25(1):387. doi: 10.1186/s12871-025-03224-6. PMID 40745279